CLINICAL TRIAL: NCT06590558
Title: Phase I/Ib Study of Eribulin in Combination With ASTX660 (Tolinapant) in Metastatic Triple Negative Breast Cancer (TNBC)
Brief Title: Testing the Addition of an Investigational Anti-Cancer Drug, ASTX660 (Tolinapant), to a Usual Chemotherapy Treatment (Eribulin) for Treatment of Advanced Triple Negative Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Manually added per CS0177524- Weekly CTEP status report.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-05666; NCI-2024-05666 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10647 (Other: Ohio State University Comprehensive Cancer Center LAO); 10647 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Invasive Breast Carcinoma; Locally Advanced HER2-Negative Breast Carcinoma; Locally Advanced Hormone Receptor-Positive Breast Carcinoma; Locally Advanced Triple-Negative Breast Carcinoma; Metastatic HER2-Negative Breast Carcinoma; Metastatic Hormone Receptor-Positive Breast Carcinoma; Metastatic Triple-Negative Breast Carcinoma; Unresectable HER2-Negative Breast Carcinoma; Unresectable Hormone Receptor-Positive Breast Carcinoma; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; eribulin; Magnetic Resonance Spectroscopy; ASTX-660; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tolinapant, eribulin) (Experimental): Patients receive tolinapant PO QD on days 1-7 and 15-21 and eribulin IV over 2-5 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, tissue biopsy, chest X-ray, and CT or MRI throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Eribulin Mesylate; Procedure: Magnetic Resonance Imaging; Drug: Tolinapant; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526 Mesylate; Halaven; Halichondrin B Analog
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Tolinapant — Given PO
  Other Names: ASTX 660; ASTX660; XIAP/cIAP1 Antagonist ASTX660
Procedure: X-Ray Imaging — Undergo chest X-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I/Ib trial tests the safety, side effects, best dose, and effectiveness of ASTX660 (tolinapant) in combination with eribulin mesylate (eribulin) in treating patients with triple negative breast cancer that cannot be removed by surgery (unresectable) or that has spread to nearby tissues or lymph nodes (locally advanced) or to other places in the body (metastatic). Tolinapant may stop the growth of tumor cells by blocking proteins, such as XIAP and cIAP1, needed for tumor cell survival. Chemotherapy drugs, such as eribulin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving tolinapant in combination with eribulin may be safe, tolerable, and/or effective in treating patients with unresectable, locally advanced, or metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of ASTX660 (tolinapant) in combination with eribulin in patients with metastatic breast cancer.

II. Determine the maximum tolerated dose (MTD) of ASTX660 (tolinapant) in combination with eribulin.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. Determine the pharmacokinetic parameters of ASTX660 (tolinapant) and eribulin when used in combination.

III. Determine the pharmacodynamic parameters of antitumor activity of ASTX660 (tolinapant) and eribulin combination.

EXPLORATORY OBJECTIVES:

I. Develop biomarkers predictive of response and resistance to ASTX660 (tolinapant) in combination with eribulin in metastatic triple negative breast cancer.

II. Investigate biomarkers and mechanisms of primary and secondary resistance to ASTX660 (tolinapant) in combination with eribulin in metastatic triple negative breast cancer.

OUTLINE: This is a dose-escalation study of tolinapant in combination with eribulin followed by a dose-expansion study.

Patients receive tolinapant orally (PO) once daily (QD) on days 1-7 and 15-21 and eribulin intravenously (IV) over 2-5 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, tissue biopsy, chest X-ray, and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast carcinoma.

  * We limit the molecular subtype to triple negative (TNBC) and hormone receptor-low and Her2 negative (hormone receptor [HR]-low/Her2[-]) breast cancer. TNBC is defined as: HER2 expression 0 or 1+ on immunohistochemistry (IHC) or non-amplified (defined as HER2/CEP17 ratio < 2 or copy number < 6) on fluorescence in situ hybridization (FISH). If HER2 expression is 2+ on IHC, negative HER2 expression must be confirmed by FISH. Pathologic diagnosis of TNBC (negative HER2 status by cytogenetics, < 1% of cells stained positive for estrogen receptor [ER] by IHC, and < 1% of cells stained positive for progesterone receptor [PR] by IHC) (Allison et al., 2020, Wolff et al., 2013). HR-low/Her2(-) is defined as: HER2 expression 0 or 1+ on IHC or non-amplified (defined as HER2/CEP17 ratio < 2 or copy number < 6) on fluorescence in situ hybridization (FISH). If HER2 expression is 2+ on IHC, negative HER2 expression must be confirmed by FISH. 1-10% of cells stained positive for ER by IHC, and/or 1-10% of cells stained positive for PR by IHC) (Allison et al., 2020, Wolff et al., 2013)
* Patients must have confirmed locally advanced and unresectable or metastatic disease by either imaging or tissue diagnosis
* Patients must have received at least 2 lines of systemic treatment for metastatic disease
* Patients must have measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) criteria
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of ASTX660 (tolinapant) in combination with eribulin mesylate in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.8 mg/dL
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional upper limit of normal (ULN) or ≤ 5 x institutional ULN if known liver metastases
* Alkaline phosphatase ≤ 3 x institutional ULN or ≤ 5 x institutional ULN if known liver and/or skeletal metastases
* Lipase ≤ 1.5 x ULN
* Creatinine ≤ 1.5 x institutional ULN OR glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2
* International normalized ratio (INR) ≤ 1.5 x ULN
* Partial thromboplastin time (PTT) ≤ 1.5 x ULN
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial provided they are on a stable regimen of anti-retroviral therapy (ART) with no medications otherwise prohibited by this protocol (e.g., drug-drug interactions)
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after central nervous system (CNS)-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better. Patients with history of known congestive heart failure (left ventricular ejection fraction [LVEF] < 50%) must have documented LVEF ≥ 50% within 12 months of study enrollment
* Patients with history of known type I or type II diabetes must have a fasting glucose level of < 120 mg/dL on at least 2 separate occasions or glycosylated hemoglobin (HbA1c) < 8.5% at screening within 14 days prior to registration
* Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that their medication dose and INR/PTT is stable
* Prophylactic antiemetics may be administered according to standard practice. The routine use of standard antiemetics, including 5-HT3 blockers, such as granisetron, ondansetron, or an equivalent agent, is allowed as needed, as long as corrected QT (QTc) interval on baseline electrocardiogram (ECG) < 480 msec
* Patients must be willing to have biopsies for this study in order to be enrolled in the dose expansion
* The effects of ASTX660 (tolinapant) on the developing human fetus are unknown. For this reason and because dual IAP antagonist agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to practice 1 highly effective contraceptive measure of birth control (with a failure rate of < 1% per year; preferably with low user dependency) during the study and for 6 months after the last dose of study treatment and must agree not to become pregnant for 6 months after completing treatment. Men with female partners of childbearing potential must agree to use a condom and advise their partners to practice 1 highly effective contraceptive measure of birth control (user dependent or with low user dependency) during the study and for at least 3 months after completing treatment, and must agree not to father a child while receiving study treatment and for at least 3 months after completing treatment
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents or concurrent anticancer therapy
* Patients who have had prior treatment with eribulin mesylate
* Patients with pre-existing neuropathy of grade 2 or higher
* Myeloid growth factors within 7 days prior to treatment start
* Platelet transfusion within 7 days prior to treatment start
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ASTX660 (tolinapant) or other agents used in study
* Immunosuppressive therapy is not allowed while on study
* Systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not permitted while on study. Previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days prior to the CT/MRI screening. If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose before the screening. Patients may be using topical or inhaled corticosteroids. Short-term (up to 7 days) systemic corticosteroids above 15 mg prednisolone or equivalent will be allowed for the management of acute conditions (e.g., treatment non-infectious pneumonitis)
* Patients with non-healing wound, ulcer, or bone fracture. Patients with compression or pathologic fractures that are stable in the opinion of the investigator may be enrolled, as long as the bone fracture is not felt to pose a high likelihood of treatment delay or difficulties in treatment adherence as per the judgement of the investigator
* Patients with active, clinically serious infections > grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] version [v]5.0) (viral, bacterial or fungal infection)
* History of known pneumocystis jiroveci pneumonia (PJP) infection or documented non-infectious pneumonitis/interstitial lung disease (ILD)
* Patients with arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
* Uncontrolled hypertension (defined as blood pressure ≥ 150/90 mm/Hg) despite optimal medical management (per investigator's opinion)
* Proteinuria as estimated by urine protein/creatinine ratio > 3.5 g/g on random urine sample or grade ≥ 3 as assessed by 24-hour urine protein collection
* Patients with history of, or current uncontrolled autoimmune disease. Patients who have adrenal or pituitary insufficiency who are stable on replacement therapy (i.e., thyroxine or physiologic corticosteroid replacement therapy that meets concomitant medication restrictions) are allowed
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because ASTX660 (tolinapant) and eribulin mesylate are anti-cancer agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ASTX660 (tolinapant) and eribulin mesylate, breastfeeding should be discontinued until 2 weeks after the mother's last dose of study drugs
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* Patients with congenital long QT syndrome, bradyarrhythmias, or taking drugs known to prolong the QT interval
* Patients unable to stop using any medication which is a moderate or strong CYP3A4 inhibitor or inducer within 2 weeks of the start of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 3 months after last dose of study drug
  Medical Dictionary for Regulatory Activities (MedDRA) terms will be used to characterized AEs which will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Descriptive statistics will be used to report the frequency according to severity of the AEs.
Dose-limiting toxicities (DLT) | Up to 4 weeks following the first administration (cycle 1 day 1) of the investigational therapy
  MedDRA terms will be used to characterized the AEs which will be graded according to the NCI CTCAE v5.0. Descriptive statistics will be used to report the frequency according to the severity of the AEs.
Maximum tolerated dose (MTD) | Up to 4 weeks
  The MTD will be defined as the highest dose at which 0 out of first 3 or 1 out of total of 6 patients experience a DLT during the first cycle of therapy, collectively 4 weeks of the investigational therapy.

SECONDARY OUTCOMES:
Overall response rate (ORR) | At start of treatment until disease progression/recurrent, assessed up to 3 years
  The best ORR is the best response recorded from the start of the treatment until disease progression/recurrence. Will be estimated along with two-sided 95% confidence intervals with the exact method of Clopper-Pearson intervals for all evaluable patients who received the investigational therapy as well as for all evaluable patients who received the investigational therapy at the MTD.
Duration of response (DOR) | At complete response (CR) or partial response (PR) to recurrent or progressive disease, assessed up to 3 years
  DOR will be measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. DOR will be analyzed using the Kaplan-Meier method.
Progression-free survival (PFS) | At start of treatment to progression or death, assessed up to 3 years
  PFS will be defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. PFS will be analyzed using the Kaplan-Meier method.
Overall survival (OS) | At start of treatment to death, assessed up to 3 years
  OS will be defined as the duration of time from start of treatment to time of death of any cause. OS will be analyzed using the Kaplan-Meier method.
Maximum concentration (Cmax) of ASTX660 (tolinapant) and eribulin | Up to day 8
  Cmax will be derived from the measured concentrations of eribulin and tolinapant by performing noncompartmental analysis or pharmacometrics. Descriptive statistics will be used to report pharmacokinetics.
Time of maximum concentration (Tmax) of ASTX660 (tolinapant) and eribulin | Up to day 8
  Tmax will be derived from the measured concentrations of eribulin and tolinapant by performing noncompartmental analysis or pharmacometrics. Descriptive statistics will be used to report pharmacokinetics.
Area under the curve (AUC) of ASTX660 (tolinapant) and eribulin | Up to day 8
  AUC will be derived from the measured concentrations of eribulin and tolinapant by performing noncompartmental analysis or pharmacometrics. Descriptive statistics will be used to report pharmacokinetics.
Half Tmax (T½) of ASTX660 (tolinapant) and eribulin | Up to day 8
  T½ will be derived from the measured concentrations of eribulin and tolinapant by performing noncompartmental analysis or pharmacometrics. Descriptive statistics will be used to report pharmacokinetics.
Clearance of ASTX660 (tolinapant) and eribulin | Up to day 8
  Clearance will be derived from the measured concentrations of eribulin and tolinapant by performing noncompartmental analysis or pharmacometrics. Descriptive statistics will be used to report pharmacokinetics.
Change in cleaved caspase 3 levels | At pre-study and at week 5
  Change in cleaved caspase 3 levels assessed in an apoptosis multiplex immunoassay on a Luminex platform in paired pre- and on-treatment tumor biopsies. The measured levels of caspase 3 in paired pre- and on-treatment biopsies will be compared using a nonparametric paired t-test.

OTHER OUTCOMES:
Positive and negative predictive value of RIPK1 and RIPK1 in pretreatment tumor biopsies in predicting response to the investigational therapy | At pre-study and up to 3 years
Sensitivity and specificity of RIPK1 and RIPK1 in pretreatment tumor biopsies in predicting response to the investigational therapy | At pre-study and up to 3 years
Area under the receiver operating characteristic curve of RIPK1 and RIPK1 in pretreatment tumor biopsies in predicting response to the investigational therapy | At pre-study and up to 3 years
Relationship between tumor transcriptional profiles | At pre-study and at week 5
Induction of apoptosis | Up to 3 years
Epithelial-to-mesenchymal transition markers | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelley, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm